CLINICAL TRIAL: NCT00262457
Title: BIONs, for Improved Tissue Health and Pressure Sore Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was found that the devices were not suitable for the application.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3259-R
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Pressure Ulcers; Spinal Cord Injury
Keywords: electrical stimulation; Pressure Ulcers; Spinal Cord Injury
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Device: Implanted gluteal electrical stimulation system

INTERVENTIONS:
Device: Implanted gluteal electrical stimulation system — Implanted electrical stimulation system incorporating BION microstimulators

SUMMARY:
The purpose of this study was to determine the feasibility of an implanted electrical stimulation system incorporating BION microstimulators for long term use to prevent tissue breakdown in high risk patients.

DETAILED DESCRIPTION:
The overall goal of this project was to implement the use of a gluteal stimulation system incorporating BION microstimulators for pressure ulcer prevention in patients at high risk of tissue breakdown as a standard clinical practice.The specific goal of this study is to establish the feasibility of a system incorporating BION microstimulators for long term use. This will be achieved by a two phase study. The initial phase of the study will employ biomechanical testing and in-vitro evaluations to address issues of safety and system design. The specific tasks to be achieved in the initial phase are:

Biomechanical testing to characterize the device response to traumatic loading conditions.

In-vitro testing to determine the optimal configuration of the system, specifically the effects of BION orientation and placement relative to the coil.

A series of cadaveric studies to determine guidelines for the BION implantation procedure required to achieve optimal function of the gluteal stimulation system.

The second phase of the study will be a pilot clinical trail of veterans with reduced mobility in order to establish clinical utility. A two-arm crossover study of wheelchair users will be carried out. A total of 10 subjects will be recruited to the study. Participants will be randomly assigned to Group A or Group B. All subjects will receive BION microstimulators implanted bilaterally adjacent to the motor point of the gluteus maximus. Two stimulation regimes will be employed; conditioning stimulation will be applied at night to increase muscle strength and fatigue resistance of the stimulated muscles while dynamic stimulation will be employed during the day in order to facilitate regular weight shifting, thus varying seated posture and pressure distributions at the seating interface. Subjects in Group A will start using dynamic and conditioning stimulation concurrently for 6 months following implantation. They will then cease using all stimulation for a further 6 months of participation in the study. Group B will not activate their stimulation systems for 6 months following implantation. They will then commence using dynamic and conditioning stimulation for 6 months.

All subjects will be followed for a 12 month period following implantation. Tissue health assessments will be carried out at three month intervals throughout their participation in the study. Progressive changes in gluteal tissue health will assessed by:

1. Transcutaneous oxygen measurement to measure tissue blood flow.
2. Interface pressure measurement to determine pressure distribution changes over the long-term (due to muscle changes) and over the short-term (due to muscle contractions).
3. Computerized tomography (CT) to measure muscle thickness. The results of this study will provide the pilot data for the development of a full-scale clinical trial of the gluteal BION system.

ELIGIBILITY:
Inclusion Criteria:

* Motor and sensory complete spinal cord injury above the level T12.
* No open skin problems or hospitalizations during the three months prior to entrance into the study.

Exclusion Criteria:

* Age less than 18 years.
* Less than two years post-injury or loss of independent walking ability.
* More than three urinary tract infections in the previous year.
* Significant active systemic disease, e.g. heart disease, renal failure, diabetes.
* Abnormal nutritional status based on albumin and total protein levels at recruitment (3.0 for albumin, 6.0 for total protein).
* Osteomyelitis of the pelvic region, indicated by positive pelvic inlet X-ray from routine annual urologic examination or bone scan.
* Previous surgery in the perineal region that radically alters the basic anatomy, particularly regional innervation and blood supply, e.g. amputation, hemipelvectomy.
* Extensive lower motor neuron damage to motor nerves innervating the gluteal muscles or electrical excitability of gluteal muscles with lower motor neuron innervation insufficient to produce desired level of contraction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Improvement of tissue health | Not feasible

CONTACTS AND LOCATIONS:
Overall Officials: Kath M. Bogie, PhD, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States

REFERENCES:
- See also: Click here for more information about this study: BIONs, for Improved Tissue Health and Pressure Sore Prevention — http://fescenter.org/index.php?option=com_content&view=article&id=14&Itemid=36